CLINICAL TRIAL: NCT03567564
Title: Abdominal Muscle Thickness in Mechanically Ventilated Patients During Spontaneous Breathing Trials
Brief Title: Abdominal Muscle Thickness in Mechanically Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Piva Simone, Dr. Piva Simone, M.D., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: Abdominals
Record Dates: First submitted 2018-06-02; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Muscle Weakness; Weaning Failure
Keywords: abdominal muscles; spontaneous breathing trial; critically ill patients
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mechanically ventilated patients: Abdominal muscles ultrasound
  Interventions: Diagnostic Test: Abdominal muscles ultrasound

INTERVENTIONS:
Diagnostic Test: Abdominal muscles ultrasound — Abdominal muscles ultrasound during a spontaneous breathing trial using the M-mode to calculate the thickening fraction of the anterior and lateral abdominal muscles under multiple circumstances (tasks performed by the patients)

SUMMARY:
The purpose of the study is to determine to what extent the abdominal muscles contribute to airway pressure, in order to investigate the correlation between muscles weakness and extubation outcome in mechanically ventilated patients. In addition the reliability of the sonographic measurements will be assessed.

DETAILED DESCRIPTION:
The purpose of the study is to determine to what extent the abdominal muscles contribute to airway pressure, in order to investigate the correlation between muscles weakness and extubation outcome in mechanically ventilated patients. In addition the reliability of the sonographic measurements will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years old
* Patients requiring invasive mechanical ventilation including patients with endotracheal tube and tracheotomies

Exclusion Criteria:

* Patients with a previously diagnosed neuromuscular disorder (acute or chronic)
* Behavioural agitation
* Patients who are not awake and cooperative
* Previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Mechanically ventilated in ICU
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-12-28 (Estimated)

PRIMARY OUTCOMES:
Correlation between thickening fraction and SBT outcome | Measurements will be performed before SBT
  Correlation between thickening fraction of each muscles evaluated by ultrasound before the SBT and the SBT outcome.

SECONDARY OUTCOMES:
Correlation between the pressures generated by respiratory muscles and SBT outcome | Measurements will be performed before SBT
  Correlation between the pressures generated by respiratory muscles during the ultrasound measurements (Twice Transdiaphragmatic pressure, TwPdi; maximal inspiratory pressure, MIP) and SBT outcome
Inter-rater agreement | Measurements will be performed before SBT
  Concordance of measurements of abdominal muscle thickness and thickening fraction in mechanically ventilated patients performed by two different observers will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Piva, M.D., Study Director — University Of Brescia, Spedali Civili di Brescia; Ewan Goligher, M.D., Principal Investigator — University of Toronto
Locations (2):
- Toronto General Hospital Research Institute, Toronto, Canada
- Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schreiber AF, Bertoni M, Coiffard B, Fard S, Wong J, Reid WD, Brochard LJ, Piva S, Goligher EC. Abdominal Muscle Use During Spontaneous Breathing and Cough in Patients Who Are Mechanically Ventilated: A Bi-center Ultrasound Study. Chest. 2021 Oct;160(4):1316-1325. doi: 10.1016/j.chest.2021.05.053. Epub 2021 Jun 6. PMID 34090872